CLINICAL TRIAL: NCT04079569
Title: Empower Korean Families to End Tobacco Use & Smoking Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Korean Community Center of the East Bay (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TRDRP 26IP-0037
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Smoking Cessation; Lifestyle Risk Reduction
Keywords: tobacco; smoking cessation; Asian Americans
MeSH Terms: conditions — Smoking Cessation; Risk Reduction Behavior | interventions — Tobacco Products

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tobacco (Experimental): Participants will receive education delivered by a lay health worker on "Quit Smoking For a Healthy Family." Participants will receive written information on nutrition and physical activity.
  Interventions: Behavioral: Tobacco
- Healthy Living (Active Comparator): In this comparison arm, participants will receive education delivered by the lay health worker about "Healthy Living" focusing on nutrition and physical activity education. Participants will also receive the Smoking Cessation Resource Handout.
  Interventions: Behavioral: Healthy Living

INTERVENTIONS:
Behavioral: Tobacco — Quit Smoking For a Healthy Family - This is a family-based psycho-education intervention using lay health worker (LHW) outreach. LHW will be trained to recruit smoke-family dyads and provide education and information about tobacco and health, and smoking cessation resources through 2 small-group education sessions and 2 individual phone calls over a 2-month period.
  Arms: Tobacco
Behavioral: Healthy Living — In this comparison arm, participants will receive the same number of contacts on the same schedule and in the same format (2 small group sessions and 2 telephone calls). The comparison LHWs will receive training about "Healthy Living" focusing on nutrition and physical activity education. Participants will also receive the Smoking Cessation Resource Handout.
  Arms: Healthy Living

SUMMARY:
The goals of the study are to develop a culturally and linguistically appropriate intervention to promote smoking cessation and reduce secondhand smoke exposure for Korean Americans using a family-based intervention approach targeting Korean Americans ages 18 and above in the greater San Francisco Bay Area, CA, and to evaluate efficacy of the proposed intervention. The study is a randomized control trial targeting a total of 8 lay health workers (LHW) and 48 dyads of a daily smoker and a partner who will attend intervention sessions together. The research question is: Can a family-based lay health worker outreach intervention promote smoking cessation and reduce SHS exposure among Korean Americans?

ELIGIBILITY:
Inclusion Criteria:

* reside in California, United States
* for the smoker participants, they must have smoked at least 1 cigarette in the past 30 days, and have smoked either at least 1 cigarette and/or used e-cigarettes in the past 7 days, and self-identified as Korean or Korean American
* for partner participants, they must be willing to attend intervention session together with a smoker participant
* provide a valid contact telephone number and email address for pre- and post-intervention assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Abstinence | 3 months
  Biochemically verified 7-day point prevalence of cigarette abstinence at 3-month post baseline assessment (initiation of intervention)
Secondhand smoke (SHS) exposure of non-smokers | 3 months
  Biochemically verified 7-day point prevalence of SHS exposure at 3-month post baseline assessment (initiation of intervention)
Percent attendance | 3-month
  Percent of participants who attend at least 3 out of 4 planned contacts
Percentage of participants who rate the intervention as helpful | 3 months
  Participants will rate their perception as to whether or not they found the intervention to be helpful at the 3 month assessment

SECONDARY OUTCOMES:
Number of Quit attempts | 3 months
  Self-report number participants making a quit attempt(s) that lasted at least for 24 hours since baseline

CONTACTS AND LOCATIONS:
Overall Officials: Janice Y Tsoh, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Korean Community Center of the East Bay, San Leandro, California, United States

IPD SHARING:
Plan to Share IPD: No